CLINICAL TRIAL: NCT03438279
Title: Projecting Survival for Patients Treated With First-Line Ipilimumab-Nivolumab Combination Therapy Using a Prognostic Model and Cost Per Responder Model of Ipilimumab-Nivolumab Combination Therapy
Brief Title: Survival Study for Participants Treated With Ipilimumab-Nivolumab Combination Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-437
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First-Line Ipilimumab: patients who received ipilimumab as their first-line treatment
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study will review published trial literature and documents for Overall Survival (OS) to evaluate the association between the hazard of death and each baseline variable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melanoma

Exclusion Criteria:

* Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual patient data (IPD) from the ipilimumab pooled analysis of clinical trials and observational studies will be used to construct the prognostic model for OS in advanced melanoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Prognostic Model of Overall Survival (OS) | 10 years
  The OS prognostic model uses Individual patient data from a pooled analysis of 12 ipilimumab studies.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Boston, Massachusetts, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx